CLINICAL TRIAL: NCT06806943
Title: How Avatar Can Enhance Autobiographical Memory of Patients With Substance Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Le.L.A.T. Lega Lotta Aids E Tossicodipendenza (Other)
Collaborators: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Fabio Frisone, Clinical Professor, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MEM-AV
Record Dates: First submitted 2025-01-27; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Substance Use Disorder (SUD)
Keywords: autobiographical memory; substance use disorder
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: within-subject design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avatar / Face-to-face (Experimental): SUD patients were investigated using the Autobiographical Memory Test in two conditions: face-to-face and avatar-based interactions. Patients had to recall 6 neutral cue words and 6 substance-related cue words for each condition.
  Interventions: Device: avatar-based interactions

INTERVENTIONS:
Device: avatar-based interactions — SUD patients were investigated using the Autobiographical Memory Test in two conditions: face-to-face and avatar-based interactions. Patients had to recall 6 neutral cue words and 6 substance-related cue words for each condition.

SUMMARY:
The goal of this study is to investigate whether the use of artificial intelligence platforms can promote the retrieval of specific positive autobiographical memories.

DETAILED DESCRIPTION:
The decision to focus on the retrieval of positive autobiographical memories was made for ethical reasons and is not tied to any specific research hypothesis. Specifically, the study aims to assess whether artificial intelligence facilitates the sharing of personal experiences and reflection on autobiographical memories related to substance use disorders, taking into account the potential influence of individual characteristics such as recent mood state, and overall memory functioning.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of substance use disorder
* Admitted to the drug rehabilitation center for at least 3 months
* Aged 18 years or older

Exclusion Criteria:

* Previous neurological pathologies
* Previous cognitive deficits

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 42 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Change in Specific Autobiographical Memory Recall | During the intervention sessions for both conditions (avatar-based and face-to-face). This outcome directly reflects the study's objective by quantifying the change of AM recall through avatar-based interventions.
  The primary outcome measure is the difference in the number of specific autobiographical memories recalled between the avatar-based interaction condition and the face-to-face condition, as assessed by the Autobiographical Memory Test (AMT). Specificity of recalled memories are scored using standardized criteria. This measure evaluates the effectiveness of avatar-based interventions in changing AM recall in patients with substance use disorder (SUD).

SECONDARY OUTCOMES:
Latency of Autobiographical Memory Recall | During the intervention sessions for both conditions (avatar-based and face-to-face).
  The secondary outcome measure is the comparison of latency times (time taken to recall a memory) between the avatar-based interaction condition and the face-to-face condition, as recorded during the Autobiographical Memory Test (AMT). This measure evaluates whether the use of avatar-based interventions change the speed of autobiographical memory recall in patients with substance use disorder (SUD).
Pleasantness of Autobiographical Memories Recalled | During the intervention sessions for both conditions (avatar-based and face-to-face).
  The secondary outcome measure is the comparison of pleasantness ratings of autobiographical memories recalled between the avatar-based interaction condition and the face-to-face condition. Pleasantness is assessed during the Autobiographical Memory Test (AMT). This measure evaluates whether avatar-based interventions change the emotional valence of the memories retrieved by patients with substance use disorder (SUD).
Change in Age Memory Recall | During the intervention sessions for both conditions (avatar-based and face-to-face).
  The secondary outcome measure is the change in age memory recall, defined as the participants' ability to identify the age at which autobiographical memories occurred, comparing the avatar-based interaction condition to the face-to-face condition. Age memory is assessed during the Autobiographical Memory Test (AMT) for each recalled memory. This measure evaluates whether avatar-based interventions change temporal specificity in autobiographical memory recall among patients with substance use disorder (SUD).

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Frisone, PhD, Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- Le.L.A.T. Lega Lotta Aids E Tossicodipendenza, Messina, Italy

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the Individual Participant Data (IPD) starting from January 25, 2025. The data will be made available for research purposes to qualified researchers who submit a formal request and have an approved data-sharing agreement. Access will be contingent upon ensuring that proper data protection and confidentiality measures are followed, in compliance with ethical guidelines and applicable data protection laws. The data will not be shared for commercial purposes without further approval. The IPD will be made available for 5 years from the date of release.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available starting from January 25, 2025. The data will remain available for 5 years from the date of release. Access to the data will be granted to qualified researchers upon request and following approval of a data-sharing agreement to ensure proper use and confidentiality.
Access Criteria: Access to the data will be granted to qualified researchers who have a legitimate research purpose. Researchers must submit a formal request detailing the proposed study, its objectives, and the intended use of the data. Access will be contingent upon approval of a data-sharing agreement, which will outline the terms and conditions of use, including confidentiality and data security measures. The data will be provided only for research purposes and cannot be used for commercial purposes without further agreement.
URL: https://zenodo.org/me/uploads?q=&l=list&p=1&s=10&sort=newest

REFERENCES:
- [Background] Nandrino JL, Gandolphe MC, El Haj M. Autobiographical memory compromise in individuals with alcohol use disorders: Towards implications for psychotherapy research. Drug Alcohol Depend. 2017 Oct 1;179:61-70. doi: 10.1016/j.drugalcdep.2017.06.027. Epub 2017 Jul 21. PMID 28756101
- [Background] Nandrino JL, Gandolphe MC. Characterization of Self-Defining Memories in Individuals with Severe Alcohol Use Disorders After Mid-Term Abstinence: The Impact of the Emotional Valence of Memories. Alcohol Clin Exp Res. 2017 Aug;41(8):1484-1491. doi: 10.1111/acer.13424. Epub 2017 Jun 14. PMID 28556207
- [Background] De Groote C, Cottencin O, Tison P, Triquet C, Nandrino JL. Autobiographical memories cued by self-statements in patients with alcohol use disorder: linking self-conceptions to past events. Memory. 2023 May;31(5):732-746. doi: 10.1080/09658211.2023.2191899. Epub 2023 Mar 22. PMID 36950753
- [Background] Nandrino JL, El Haj M, Torre J, Naye D, Douchet H, Danel T, Cottencin O. Autobiographical Memory Deficits in Alcohol-Dependent Patients with Short- and Long-Term Abstinence. Alcohol Clin Exp Res. 2016 Apr;40(4):865-73. doi: 10.1111/acer.13001. Epub 2016 Mar 17. PMID 26990362
- [Background] Fernandez-Alvarez J, Colombo D, Suso-Ribera C, Chirico A, Serino S, Di Lernia D, Palacios AG, Riva G, Botella C. Using virtual reality to target positive autobiographical memory in individuals with moderate-to-moderately severe depressive symptoms: A single case experimental design. Internet Interv. 2021 May 27;25:100407. doi: 10.1016/j.invent.2021.100407. eCollection 2021 Sep. PMID 34401366
- [Background] Lenormand D, Mentec I, Gaston-Bellegarde A, Orriols E, Piolino P. Decoding episodic autobiographical memory in naturalistic virtual reality. Sci Rep. 2024 Oct 27;14(1):25639. doi: 10.1038/s41598-024-76944-3. PMID 39463396
- [Background] Frisone F, Brizzi G, Riva G. VR-MEM: Harnessing Virtual Reality for Autobiographical Memory Enhancement in High School Settings. Cyberpsychol Behav Soc Netw. 2024 Jan;27(1):91-93. doi: 10.1089/cyber.2023.29300.ceu. Epub 2023 Nov 16. No abstract available. PMID 37972046
- [Background] Frisone F, Calabro G, Rossi C, Riva G. MEM-AV: A VR-Based Approach to Improve Autobiographical Memory Retrieval in Addiction. Cyberpsychol Behav Soc Netw. 2024 May;27(5):353-355. doi: 10.1089/cyber.2024.42624. Epub 2024 May 8. No abstract available. PMID 38717129
- [Background] Pitel AL, Eustache F, Beaunieux H. Component processes of memory in alcoholism: pattern of compromise and neural substrates. Handb Clin Neurol. 2014;125:211-25. doi: 10.1016/B978-0-444-62619-6.00013-6. PMID 25307577
- [Background] Conway MA, Pleydell-Pearce CW. The construction of autobiographical memories in the self-memory system. Psychol Rev. 2000 Apr;107(2):261-88. doi: 10.1037/0033-295x.107.2.261. PMID 10789197